CLINICAL TRIAL: NCT03447873
Title: Is Dual Therapy as Effective as Triple Therapy Regarding CD4+/CD8+ Ratio Recovery and Improvement of Immune Activation and Inflammation in HIV-infected Patients With Consistent Plasma Viral Load Suppression (Tridual)
Brief Title: Tripe Versus Dual Antiretroviral Therapy in HIV-infected Patients With Virological Suppression (Tridual)
Acronym: Tridual
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Luis F. Lopez-Cortes, Senior Researcher Andalusian Health System, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIS-TAR-01-2016; 2016-005226-11 (EudraCT Number)
Record Dates: First submitted 2017-07-11; First posted 2018-02-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: HIV Infections
Keywords: Antiretroviral treatment; Treatment simplification; Dual therapy; Immune recovery
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple therapy (Active Comparator): To Continue with triple therapy with Elvitegravir/cobicistat + tenofovir alafenamide + emtricitabine or Dolutegravir + abacavir + lamivudine once daily.
  Interventions: Drug: Continue with triple therapy
- Switch to dual therapy A (Experimental): Switch to dual therapy with Darunavir/cobicistat (800150 mg) + lamivudine (300 mg) once daily once daily.
  Interventions: Drug: Switch to DTG + 3TC
- Switch to dual therapy B (Experimental): Switch to dual therapy with Dolutegravir (50 mg) + lamivudine (300 mg) once daily
  Interventions: Drug: Switch to DRV/cobicistat + 3TC

INTERVENTIONS:
Drug: Continue with triple therapy — To continue with triple therapy
  Arms: Triple therapy
Drug: Switch to DTG + 3TC — Switch to dolutegravir + lamivudine once daily
  Arms: Switch to dual therapy A
Drug: Switch to DRV/cobicistat + 3TC — Switch to darunavir/cobicistat + lamivudine once daily
  Arms: Switch to dual therapy B

SUMMARY:
The persistence of an aberrant state of immune activation and inflammation (pIA) may contribute to the emergence of serious non-AIDS events which carry a higher morbimortality in HIV-infected patients. Although combined antiretroviral treatment (cART) reduces both cellular and soluble activation markers, it fails to completely control pIA despite consistent plasma viral load suppression. One of the mechanisms involved in pIA is may be an incomplete suppression of viral replication not reflected by plasma viral load, which only reflects a balance between viral replication and clearance of HIV-RNA. In addition, low-level viremia detected in most HIV-1-infected patients despite years on cART. Unintegrated 2-LTR HIV-DNA, and cellular associated HIV-RNAs, as products of active integrated DNA transcription, support this issue.

Furthermore, the key rationales behind simplifying cART are a reduction of toxicities, lower risk of resistance mutations in case of virological failure and saving costs. One of these simplification strategies is a dual therapy which, based on the data up to date and in our clinical experience, has similar virological efficacy than cART. However, it is unknown if this strategy could increase the persistent HIV-1 replication and, therefore, pIA. The CD4+/CD8+ T cell ratio as a marker of immune recovery, the changes in T cell immune activation, senescence, exhaustion and apoptosis, and the cellular associated HIV-DNA and -RNA would answer the question if simplification to dual therapy would provide less control of residual HIV replication and, therefore, a detriment on pIA compared to triple therapy and, therefore, would worsen the patients' long-term prognosis.

DETAILED DESCRIPTION:
Primary Outcome Measures: to evaluate the changes in the CD4/CD8 ratio, immune activation and other immunologic parameters at 48 weeks after switching to dual therapy based on dolutegravir plus emtricitabine o darunavir/cobicistat plus emtricitabine versus to continue on triple therapy based on integrase inhibitor plus 2 analogs Secondary Outcome Measures: to evaluate the changes in the CD4/CD8 ratio, immune activation and other immunologic parameters at 96 weeks after switching to dual therapy based on dolutegravir plus emtricitabine o darunavir/cobicistat plus emtricitabine versus to continue on triple therapy based on integrase inhibitor plus 2 analogs

Method: randomized clinical trial in which adult HIV-infected patients with an undetectable plasma HIV-RNA for at least one year on a triple therapy based on integrase inhibitors plus two nucleos(t)ide analogs will be randomized in 3 groups (1:1:1) with 4 strata according to the previous time with undetectable viral load to:

1. Continue the previous ART based on Elvitegravircobicistat 150150 mg + tenofovir alafenamide 10 mg + emtricitabine 200 mg (Genvoya™) o Dolutegravir 50 mg + abacavir 600 mg + lamivudine 300 mg (Triumeq™) once daily.

   Or to switch to:
2. Darunavir/cobicistat (800150 mg) + 3TC (300 mg) once daily or
3. Dolutegravir (50 mg) + 3TC (300 mg) once daily.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected patients ≥ 18 years of age.
* Starting date of antiretroviral treatment later than 01/01/2010
* Plasma HIV-1 RNA <20 copies/ml for at least one year on triple therapy
* Antiretroviral treatment based on an integrase inhibitor plus two nucleos(t)ide analogs in the last 6 months.
* Signed written informed consent prior to inclusion.

Exclusion Criteria:

* Primary resistance to any of the drugs included in the study.
* Active opportunistic infection.
* Pregnancy at inclusion or during the follow-up
* Active hepatitis C and/or B virus co-infection.
* Cirrhosis, portal hypertension and/or hypersplenism of any etiology.
* Current or past malignancies subsidiary of treatment with corticosteroids, immunomodulatory agents, interferon or chemotherapeutic agents.
* Any laboratory abnormality grade 3 or 4 according to the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS.
* Concomitant use of drugs with potential major interactions with the prescribed drugs according to the respective full prescribing information.
* Estimated creatinine clearance <50 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
CD4/CD8 ratio | 48 weeks
  To evaluate if a triple therapy based on integrase inhibitors plus two nucleos(t)ide analogs will provide a higher CD4+/CD8+ T cell ratio recovery compared with dual therapies based on darunavir/cobicistat plus lamivudine or dolutegravir plus lamivudine after 48 weeks of treatment in HIV-infected patients with consistent plasma viral load suppression.

SECONDARY OUTCOMES:
Immune activation | 48 weeks
  To assess whether dual therapies provide an increase in immune activation and inflammation compared to triple therapy assessed by the expression of HLA-DR and CD38 in both of CD4+ and CD8+ T cells and sCD14 after 48 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, PhD, Study Director — Virgen del Rocio University Hospital. Seville. Spain
Locations (1):
- Virgen del Rocio University Hospital, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Muela E, Trujillo-Rodriguez M, Serna-Gallego A, Saborido-Alconchel A, Ruiz-Mateos E, Lopez-Cortes LF, Gutierrez-Valencia A. HIV-1-specific T-cell responses and exhaustion profiles in people with HIV after switching to dual therapy vs. maintaining triple therapy based on integrase inhibitors. Biomed Pharmacother. 2023 Dec;168:115750. doi: 10.1016/j.biopha.2023.115750. Epub 2023 Oct 21. PMID 37871555